CLINICAL TRIAL: NCT01325662
Title: A Clinical Study to Evaluate a Modified Serial CSF Sampling Method by Indwelling Lumbar Catheter in Healthy Volunteers
Brief Title: A Study to Evaluate the Use of an Indwelling Catheter to Obtain Cerebrospinal Fluid (CSF) by Low-rate Continuous Sampling (MK-0000-211)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-211
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continuous drip sampling: Sampling at ~0.6 cc / hour (~1.2 cc / 2 hours, or lowest feasible rate given technical requirements and volume requirements for core analytes assays)
- Intermittent sampling: Sampling at 4 cc every 2 hours (+ 2 cc dead space clearance, total = 6 cc / 2 hours)

SUMMARY:
This is a study to evaluate the feasibility and tolerability of low-rate continuous Cerebrospinal Fluid (CSF) sampling and to estimate the number of participants who exhibit severe baseline instability of CSF amyloid beta isoform Aß40 concentrations in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health
* Must have a body mass index greater than or equal to 18 kg/m^2 and less than or equal to 30 kg/m^2

Exclusion Criteria:

* Is pregnant, nursing, or plans to become pregnant
* Has clinically significant cardiovascular, renal, hepatic, gastrointestinal (GI), neurological, endocrine, hematological, dermatological or metabolic disease, or clinically significant abnormalities, as determined by medical history, physical examination, electrocardiogram, vital signs, or laboratory tests
* Has a history of migraine headaches
* Has a history of recent lumbar CSF sampling within 3 weeks prior to screening, history of lumbar spine surgery, or chronic low back pain or injury
* Has an infection or inflammation of the skin in or in close proximity to the area of the lumbar puncture site
* Has a history of a seizure disorder
* Is noted to have papilledema or clinically significant focal neurological deficits at the screening physical examination, as well as abnormalities of CSF pressure on initial testing once access to the lumbar space is achieved
* Has absolute or relative anatomic abnormalities that would be a contraindication to lumbar puncture
* Is a heavy consumer of alcohol
* Has used nicotine in the past 6 months
* Has a history of a significant psychiatric disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers from general population
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Increase in CSF Aβ40 levels as measured by the new low flow continuous drip sampling method | Up to 24 hours

SECONDARY OUTCOMES:
Increase in CSF Aβ40 levels as measured by the current intermittent drip sampling method | Up to 24 hours